CLINICAL TRIAL: NCT02772744
Title: Determining the Sustained Virologic Response of Declatasvir in Egyptian Patients With Hepatitis C Virus Genotype 4
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Negida, Mr., Zagazig University
Other Study IDs: 2667-20-3-2016
Record Dates: First submitted 2016-03-24; First posted 2016-05-13 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C
Keywords: Hepatitis C virus genotype 4; Antiviral; Virologic Response
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; Tablets; Sofosbuvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1: Easy to treat group: * Treatment naïve
  * Total serum bilirubin ≤ 1.2 mg/dl
  * Serum albumin ≥ 3.5 g/dl
  * International normalized ratio ≤ 1.2
  * Platelet count ≥ 150000 mm3
  This group will be receiving Sofosbuvir + daclatasvir for 12 weeks.
  Interventions: Drug: Daclatasvir 60 MG Oral Tablet [Daklinza]; Drug: Sofosbuvir 400 MG Oral Tablet [Sovaldi]
- Group 2: Difficult to treat group: * Peg interferon treatment experienced.
  * Total serum bilirubin ≥ 1.2 mg/dl
  * Serum albumin ≤ 3.5 g/dl
  * International normalized ratio ≥ 1.2
  * Platelet count ≤ 150000 mm3
  This group will be receiving Sofosbuvir + daclatasvir + ribavirin for 12 weeks.
  Interventions: Drug: Daclatasvir 60 MG Oral Tablet [Daklinza]; Drug: Sofosbuvir 400 MG Oral Tablet [Sovaldi]; Drug: Ribavirin Oral Product
- Group 3: Sofosbuvir resistant cases: This is the group of patients who failed in previous Sofosbuvir treatment regiment. This group will be receiving Sofosbuvir + daclatasvir + ribavirin for 24 weeks.
  Interventions: Drug: Daclatasvir 60 MG Oral Tablet [Daklinza]; Drug: Sofosbuvir 400 MG Oral Tablet [Sovaldi]; Drug: Ribavirin Oral Product

INTERVENTIONS:
Drug: Daclatasvir 60 MG Oral Tablet [Daklinza] — Daclatasvir (60 MG) is a potent, pan-genotypic inhibitor of the HCV NS5A protein
Drug: Sofosbuvir 400 MG Oral Tablet [Sovaldi] — Sofosbuvir (400 MG) is a nucleotide analogue HCV NS5B polymerase inhibitor
Drug: Ribavirin Oral Product — Ribavirin (twice-daily) dosed according to body weight (<75 kg, 1000 mg daily; ≥75 kg, 1200 mg daily)
  Groups: Group 2: Difficult to treat group; Group 3: Sofosbuvir resistant cases

SUMMARY:
This is a prospective, cohort study in Faculty of Medicine, Zagazig University, Egypt. From June to December, 2016, investigators will follow up patients with chronic Hepatitis C virus genotype 4 receiving daclatasvir-sofosbuvir treatment regimen within the national program of Egyptian ministry of health and population. The primary outcomes are safety of the treatment and the sustained virologic response 12 weeks after discontinuation of therapy. For the secondary outcomes, investigators will measure the change in health related quality of life and investigate the genetic sequence of viral RNA of resistant patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCV genotype 4
* Age ≥ 18 years
* HCV RNA≥ 104 IU/mL
* Screening ECG without clinically significant abnormalities.

Exclusion Criteria:

* Total serum bilirubin > 3 mg/dl.
* Serum albumin < 2.8 g/dl.
* INR ≥ 1.7
* Platelet count < 50000/mm3.
* Hepatic cell carcinoma except four weeks after intervention aiming to cure with no evidence of activity by dynamic imaging (CT or MRI).
* Extra hepatic malignancy except after two years of disease free interval
* Pregnancy or inability to use contraception.
* Inadequately controlled diabetes mellitus (HbA1c > 9%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include male or female patients ≥ 18 years, HCV RNA≥ 104 IU/mL, HCV genotype 4, screening ECG without clinically significant abnormalities.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy measured by Sustained Virologic Response Rate | 12 weeks posttreatment
Incidence of grade 3/4 adverse events [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
Incidence of Neutropenia [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
  Neutropenia: Grade 3, 500-749/mm3; Grade 4, <500/mm3
Incidence of Lymphopenia [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
  Lymphopenia: Grade 3, 350-499/mm3; Grade 4, <350/mm3
Incidence of anaemia [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
  Anaemia: Grade 3, haemoglobin 7.0-8.9 g/dL; Grade 4, <7.0 g/dL
Incidence of Thrombocytopenia [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
  Thrombocytopenia: Grade 3, 25 000-49 999/mm3; Grade 4, <25 000/mm3
Incidence of (Increased total Bilirubin) [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
  Bilirubin elevations: Grade 3, 2.6-5×ULN; Grade 4, >5×ULN
Incidence of elevated Alanine Aminotransferase [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
  Alanine Aminotransferase elevations: Grade 3, 5.1-10×upper limit of normal (ULN); Grade 4, >10×ULN
Incidence of Fatigue [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
Incidence of Headache [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
Incidence of Pruritus [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
Incidence of Insomnia [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
Incidence of Rash [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
Incidence of Nausea [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)
Incidence of Myalgia [Safety] | Within the treatment period (12 or 24 weeks according to the treatment regimen)

SECONDARY OUTCOMES:
Health Related Quality of Life (HRQoL) | 24 weeks
  HRQoL will be assessed using the Arabic version of SF-36 questionnaire (SF-36™ Health Survey)

CONTACTS AND LOCATIONS:
Overall Officials: Samah A Loutfy, Study Director — National Cancer Institute, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jensen D, Sherman KE, Hezode C, Pol S, Zeuzem S, de Ledinghen V, Tran A, Elkhashab M, Younes ZH, Kugelmas M, Mauss S, Everson G, Luketic V, Vierling J, Serfaty L, Brunetto M, Heo J, Bernstein D, McPhee F, Hennicken D, Mendez P, Hughes E, Noviello S; HALLMARK-QUAD Study Team. Daclatasvir and asunaprevir plus peginterferon alfa and ribavirin in HCV genotype 1 or 4 non-responders. J Hepatol. 2015 Jul;63(1):30-7. doi: 10.1016/j.jhep.2015.02.018. Epub 2015 Feb 19. PMID 25703086
- [Background] Hezode C, Alric L, Brown A, Hassanein T, Rizzetto M, Buti M, Bourliere M, Thabut D, Molina E, Rustgi V, Samuel D, McPhee F, Liu Z, Yin PD, Hughes E, Treitel M; COMMAND-4 study team. Randomized controlled trial of the NS5A inhibitor daclatasvir plus pegylated interferon and ribavirin for HCV genotype-4 (COMMAND-4). Antivir Ther. 2015 Aug 27;21(3):195-205. doi: 10.3851/IMP2985. Online ahead of print. PMID 26313445
- [Background] Wyles DL, Ruane PJ, Sulkowski MS, Dieterich D, Luetkemeyer A, Morgan TR, Sherman KE, Dretler R, Fishbein D, Gathe JC Jr, Henn S, Hinestrosa F, Huynh C, McDonald C, Mills A, Overton ET, Ramgopal M, Rashbaum B, Ray G, Scarsella A, Yozviak J, McPhee F, Liu Z, Hughes E, Yin PD, Noviello S, Ackerman P; ALLY-2 Investigators. Daclatasvir plus Sofosbuvir for HCV in Patients Coinfected with HIV-1. N Engl J Med. 2015 Aug 20;373(8):714-25. doi: 10.1056/NEJMoa1503153. Epub 2015 Jul 21. PMID 26196502
- See also: Related Info — http://www.accessdata.fda.gov/drugsatfda_docs/label/2015/206843Orig1s000lbl.pdf